CLINICAL TRIAL: NCT06167902
Title: The Metabolic Effects of Ginseng Oligopeptide Preparation on Non- Alcoholic Fatty Liver Disease With Obesity: a Randomized Controlled Double-blind Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ginseng oligopeptide 1.0
Record Dates: First submitted 2023-11-29; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Asian ginseng; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ginseng oligopeptide group (Experimental)
  Interventions: Other: Ginseng oligopeptide (Ginseng extract）
- The placebo group (Placebo Comparator)
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Other: Ginseng oligopeptide (Ginseng extract） — The experimental group was given ginseng oligopeptide preparation 1.2g per day orally.
  Arms: Ginseng oligopeptide group
Other: Maltodextrin — The control group was treated with placebo maltodextrin 1.2g/d
  Arms: The placebo group

SUMMARY:
To investigate the effect of ginseng oligopeptide on nonalcoholic fatty liver disease with obesity and clarify its intervention mechanism in theory, which will contribute to the prevention and treatment of non-alcoholic fatty liver more scientifically and effectively.The patients were randomly divided into two groups. One group of patients took ginseng oligopeptide orally, and the other group took placebo. The liver function, blood lipid, blood glucose, liver B ultrasound and other indicators were observed to further determine the efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for non-alcoholic fatty liver disease ;
* Aged 18-65 years old;
* ALT, AST, GGT≤2×Upper Limit Of Normal（ULN）;
* BMI≥28Kg/㎡;
* Patients signed the relevant informed consent on a voluntary basis.

Exclusion Criteria:

* Under 18 years old and over 65 years old;
* Allergic to the ingredients of ginseng oligopeptide preparation;
* Serum ALT, AST, GGT>2ULN;
* Currently taking oral hepatoprotective drugs such as reduced glutathione, polyene phosphatidylcholine, and silibinin, etc.;
* Subjects participating in other clinical trials;
* Pregnant or lactating women;
* Complicated with serious diseases of the digestive system or other systems, such as chronic gastrointestinal diseases and chronic diseases causing digestive malabsorption,Kidney disease, hematological system or autoimmune diseases;
* Other populations that were deemed by the investigators to be ineligible for the trial may reduce or complicate enrollment patients with chemotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-25 (Estimated); Primary Completion 2024-12-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Alanine aminotransferase (ALT) | The day of enrollment, day 60 and day 120 after enrollment.
  Liver function
aspartate aminotransferase (AST) | The day of enrollment, day 60 and day 120 after enrollment.
  Liver function
glutamyltransferase (GGT). | The day of enrollment, day 60 and day 120 after enrollment.
  Liver function

IPD SHARING:
Plan to Share IPD: No